CLINICAL TRIAL: NCT06385184
Title: Social Behaviors and Quality of Life in Individuals With Parkinson's Disease
Brief Title: Social & QoL Behaviors in Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Gregory Wallace (Other)
Responsible Party: Sponsor-Investigator, Gregory Wallace, PI, George Washington University
Organization: George Washington University (Other)
Other Study IDs: NCR234859
Record Dates: First submitted 2024-04-18; First posted 2024-04-25 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Parkinson's disease: This group includes adults who:
  * Have been diagnosed with Parkinsons Disease by a healthcare professional
  * Are at least 40 years old and
  * Do not possess a diagnosis of autism or any other developmental disability (e.g., Down syndrome)
  Interventions: Other: No Intervention
- Neurotypical adults: This group includes adults who:
  * Are at least 40 years old
  * Do not have a diagnosis of Parkinsons Disease or any form of dementia and
  * Do not have a diagnosis of autism or any other developmental disability (e.g., Down syndrome)
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Observational study with no intervention

SUMMARY:
Adults with Parkinson's Disease experience an array of challenges and changes in daily living, behaviors, and functioning throughout the progression of their condition. The investigators want to learn more about the effects of Parkinson's Disease on individuals' social behavior and quality of life (QoL) compared to people of the same age without Parkinson's Disease.

ELIGIBILITY:
Parkinson's disease group

Inclusion Criteria:

* Have been diagnosed with Parkinsons Disease by a healthcare professional
* Are at least 40 years old

Exclusion Criteria:

* Possess a diagnosis of autism or any other developmental disability (e.g., Down syndrome)

Neurotypical group

Inclusion Criteria:

* Are at least 40 years old

Exclusion Criteria:

* Have been diagnosed with Parkinson's disease by a healthcare professional
* Possess a diagnosis of autism or any other developmental disability (e.g., Down syndrome)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study includes both 40+ year old adults with Parkinson's disease and 40+ year old neurotypical adults
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Subjective Quality of Life | through study completion, an average of 1 year
  satisfaction with different aspects of life, such as health and social relationships
Social Behavior | through study completion, an average of 1 year
  ability to interact with others
Activities of Daily Living | through study completion, an average of 1 year
  ability to complete tasks to be independent
Mental Health | through study completion, an average of 1 year
  depression and anxiety symptoms
Cognition | through study completion, an average of 1 year
  memory and executive function challenges and strengths

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Wallace, PhD, Principal Investigator — George Washington University
Locations (1):
- The George Washington University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Currently, there is no plan to share participant data with other researchers.